CLINICAL TRIAL: NCT02572284
Title: A Phase I Dose Escalation Study of Preoperative Stereotactic Body Radiation Therapy (SBRT) for High Risk Prostate Cancer
Brief Title: Dose Escalation Study of Preoperative SBRT for High Risk Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18201
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: Stereotactic Body Radiation Therapy (SBRT); High Risk Prostate Cancer; Preoperative SBRT; Prostate Adenocarcinoma; Prostatectomy; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Radiotherapy; Prostatectomy; Surgical Procedures, Operative; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation of SBRT (Experimental): Stereotactic Body Radiation Therapy (SBRT) followed by prostatectomy and Quality of Life questionnaires. The radiation will be given for only 5 days. Conventional radiation to the prostate is given over 7-8 weeks.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Prostatectomy; Other: Quality of Life Questionnaires

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — The first group of patients to enter the study will receive 5 Gy of SBRT per day for 5 days, the second group will receive 6 Gy per day for 5 days. Each treatment will take about 3 minutes and be given as an outpatient at Moffitt Cancer Center.
  Other Names: radiation therapy
Procedure: Prostatectomy — About 4-6 weeks after SBRT, participants will have a prostatectomy.
  Other Names: surgery
Other: Quality of Life Questionnaires — Patient assessed health-related quality of life (HRQOL). Quality of Life (QOL) will be assessed using Prostate Symptom Score (IPSS), rectal assessment scale (RAS), sexual health inventory for men (SHIM), and Expanded Prostate Cancer Index Composite (EPIC) patient questionnaires: administered prior to SBRT, and at 2 weeks, 4 weeks, 2 months and then every 3 months up to 18 months post-prostatectomy.
  Other Names: questionnaire

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad, of different doses of SBRT given before prostatectomy. Depending when participants enter the study, they will be treated with either 5 or 6 gray (Gy) per day of radiation. A Gy is a measure of radiation dose. The standard dose is 10Gy per day when SBRT is the only treatment to the prostate and no surgery is planned. The researchers want to see which dose of radiation will work best with the least amount of side effects. About 4-6 weeks after SBRT, participants will have a prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven prostate adenocarcinoma.
* Clinical stage ≤T3a based on digital rectal exam and/or ≤T3a based on MRI (if done); N0-Nx; M0-Mx (AJCC 7th Edition)
* Prostate-specific antigen (PSA) ≤ 80 ng/ml, obtained within 3 months.
* Patients belonging in the National Comprehensive Cancer Network (NCCN) high recurrence risk group. High risk: Clinical stage T3a, or Gleason score = 8-10, or PSA >20 ng/mL.
* Prostate volume: ≤ 80 cc on transrectal ultrasound
* IPSS score ≤15
* Zubrod performance status 0-2 or equivalent
* No prior total prostatectomy or cryotherapy of the prostate. Prior transurethral resection or laser ablation is permitted.
* No prior radiotherapy to the prostate or lower pelvis
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion
* No history of an invasive malignancy (other than this prostate cancer, or non-metastatic basal or squamous skin cancers) in the last 5 years
* No androgen deprivation therapy (ADT) can be prescribed prior to or during radiation therapy
* Must be able to have gold fiducial markers placed in the prostate or, if patient already has fiducial markers placed, they must be in accordance with the protocol specifications
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to fill out IPSS, SHIM, and EPIC quality of life forms
* Age ≥18 years
* IPSS (AUA) score ≤15

Exclusion Criteria:

* Does not have a diagnosis of prostate adenocarcinoma
* Has very low risk, low risk, intermediate risk or very high risk disease as defined by the NCCN
* Has stage N1 or M1 (metastatic) disease
* Has a PSA of greater than 80 ng/ml obtained no greater than 3 months prior to randomization
* Prostate volume greater than 80 cc on transrectal ultrasound
* Zubrod performance status 3 or greater
* Prior total prostatectomy or cryotherapy of the prostate
* Prior radiation therapy to the pelvis
* Implanted hardware which limits treatment planning or delivery (determined by the investigator).
* Diagnosis of an invasive malignancy within 5 years (other than current prostate cancer or non-metastatic basal or squamous skin cancers)
* The use of androgen deprivation therapy (ADT) prior to registration or during radiation
* Inability to have gold fiducial markers placed in the prostate, or fiducial markers already placed, that are not in accordance with the protocol
* Unwilling or inability to give informed consent
* Not willing to fill out IPSS, SHIM, and EPIC quality of life questionnaires
* IPSS score >15

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Up to 28 ± 5 days post-prostatectomy
  Acute dose-limiting toxicity and quality of life due to preoperative SBRT followed by robotic-assisted laparoscopic radical prostatectomy at 14 ± 5 days and 28 ± 5 days post-prostatectomy in high risk prostate cancer patients. In order to assess the toxicity of preoperative SBRT, the severity of specific events will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4 form where a score of ≥3 is considered dose-limiting.

SECONDARY OUTCOMES:
Occurrence of Late Toxicity | 90+ days after start of radiotherapy
  Late (defined as occurring more than 90 days after the start of radiotherapy) toxicity that is grade 2 or more as defined by the Common Terminology Criteria for Adverse Events version 4.
Mean Catheterization Time for Study Participants | Up to 18 months post surgery
  Mean catheterization time for study participants, compared to existing mean statistics for robotic-assisted laparoscopic radical prostatectomy.
Mean Hospital Stay for Study Participants | Up to 18 months post surgery
  Mean hospital stay for study participants, compared to existing mean statistics for robotic-assisted laparoscopic radical prostatectomy.
Reoperation Rate for Study Participants | Up to 18 months post surgery
  Mean reoperation rate for study participants, compared to existing mean statistics for robotic-assisted laparoscopic radical prostatectomy.
Patient-Assessed Changes in Health-Related Quality of Life (HRQOL) - Expanded Prostate Cancer Index Composite (EPIC) | Up to 18 months post surgery
  Administered prior to SBRT, and at 2 weeks, 4 weeks, 2 months and then every 3 months up to 18 months post-prostatectomy. The 26-item, short-form version of the Expanded Prostate Cancer Index Composite (EPIC) is a validated questionnaire used to assess HRQOL in prostate cancer patients. EPIC includes 4 domains: urinary, bowel, sexual, and hormonal. There are summary, i.e., overall, scores and function and bother subscale scores for each of the 4 domains. The urinary domain has 2 additional subscales: incontinence and irritative/obstructive. Domains and subscales are scored using a 0-100 grading system, with a higher score indicating a better quality of life.
Patient-Assessed Changes in HRQOL - International Prostate Symptom Score (IPSS) | Up to 18 months post surgery
  Administered prior to SBRT, and at 2 weeks, 4 weeks, 2 months and then every 3 months up to 18 months post-prostatectomy. The IPSS will be used to assess changes in urinary toxicity. Scoring is 0, 1, 2, 3, 4, 5 per question, Total IPSS Score out of 35 points from 7 questions. Descriptive summaries of scores at baseline and each subsequent follow up will include means and standard deviations.
Patient-Assessed Changes in HRQOL - Rectal Assessment Scale (RAS) | Up to 18 months post surgery
  Administered prior to SBRT, and at 2 weeks, 4 weeks, 2 months and then every 3 months up to 18 months post-prostatectomy. The RAS will be used to assess changes in rectal toxicity. Scoring is 0, 1, 2, 3 per question, Total RAS Score out of 15 points from 5 questions. Descriptive summaries of scores at baseline and each subsequent follow up will include means and standard deviations.
Patient-Assessed Changes in HRQOL - Sexual Health Inventory for Men (SHIM) | Up to 18 months post surgery
  Administered prior to SBRT, and at 2 weeks, 4 weeks, 2 months and then every 3 months up to 18 months post-prostatectomy. The SHIM will be used to assess changes in sexual toxicity. Scoring is 0, 1, 2, 3, 4, 5 per question, Total SHIM score out of 25 points from 5 questions. Descriptive summaries of scores at baseline and each subsequent follow up will include means and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johnstone, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Julio Pow-Sang, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/